CLINICAL TRIAL: NCT03338608
Title: Influence of Platysmal Incision on Cosmetic Satisfaction Outcomes in Anterior Cervical Spine Surgery Patients
Brief Title: Platysma Incision Cosmesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-36610
Record Dates: First submitted 2017-11-03; First posted 2017-11-09 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Wound Heal
Keywords: Cosmesis; Wound Healing; Anterior Cervical Decompression and Fusion; ACDF; Platysma
MeSH Terms: interventions — Gene Fusion

STUDY DESIGN:
Intervention Model Description: There are two groups. One group will have the vertical platysma incision and the other group will have the transverse incision.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vertical Platysma Incision (Experimental): Patients in this arm who have anterior cervical decompression and fusion will receive the vertical platysma incision.
  Interventions: Procedure: Anterior Cervical Decompression and Fusion; Procedure: Vertical Platysma Incision
- Transverse Platysma Incision (Experimental): Patients in this arm who have anterior cervical decompression and fusion will receive the transverse platysma incision.
  Interventions: Procedure: Anterior Cervical Decompression and Fusion; Procedure: Transverse Platysma Incision

INTERVENTIONS:
Procedure: Anterior Cervical Decompression and Fusion — Patients will receive the anterior cervical decompression and fusion as part of their standard of care. They will be randomized to either receive the vertical or transverse platysma incision.
Procedure: Vertical Platysma Incision — A vertical platysma Incision will be used for the anterior cervical decompression and fusion surgical procedure
  Arms: Vertical Platysma Incision
Procedure: Transverse Platysma Incision — A transverse platysma incision will be used for the anterior cervical decompression and fusion surgical procedure
  Arms: Transverse Platysma Incision

SUMMARY:
The anterior cervical fusion and decompression (ACDF) surgery provides direct access to symptomatic areas of the cervical spine. Cosmesis, including factors like wound healing, is an important issue for patients who undergo surgery on anterior neck structures. One significant factor that impacts cosmetic healing in patients who undergo the ACDF surgery is whether a vertical or transverse incision of the platysma muscle in the neck was used to access the cervical spine.

The purpose of the present study is to compare cosmetic outcomes in vertical versus transverse platysmal incisions for anterior cervical spine exposures. Researchers intend to analyze this effect with a prospective comparative study model. A targeted number of 100 patients who undergo anterior cervical surgery, as part of their standard of care, will be randomized to receive either a transverse or vertical platysmal incision during the exposure part of their procedure. Informed consent for inclusion in the study, as approved by the Institutional Review Board, will be obtained from all patients in addition to consent for the surgical procedure. Regardless of the platysmal incision, all patients will receive a standard transverse skin incision, as is done routinely in anterior cervical exposures. After the surgery, all closures will be done in a standard manner.

These patients will be followed up in the clinic at two weeks, three months, six months, and one year. They will be evaluated for wound healing and incision cosmesis using a modification of The Hollander Wound Evaluation Scale. Clinical photographs of the patients' necks will be captured during these visits in a manner that does not reveal any patient identifiers in any way. The incisions and overall cosmesis will be graded using the scale mentioned above. The data will be analyzed to determine if a transverse platysmal incision offers better cosmetic results than a vertical platysmal incision, or vice versa, and will also be used to validate the modified wound evaluation scale.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing elective Anterior Cervical Decompression and Fusion surgery for degenerative spinal pathologies by Dr. Tony Tannoury or Dr. Chadi Tannoury at Boston Medical Center as part of their standard of care.

Exclusion Criteria:

* Patients undergoing revision anterior cervical spine surgeries with a pre-existing scar. Patients with cervical spine tumors/neoplastic pathologies. Patients undergoing surgery for cervical spine trauma.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2019-09-15 (Actual); Study Completion 2019-09-15 (Actual)

PRIMARY OUTCOMES:
Modified version of the Hollander wound evaluation scale | 2 week follow up visit
  Includes several factors of cosmetic wound healing (skin puckering, patient satisfaction, etc.). Based on photographic and patient follow-up information
Modified version of the Hollander wound evaluation scale | 3 months follow up visit
  Includes several factors of cosmetic wound healing (skin puckering, patient satisfaction, etc.). Based on photographic and patient follow-up information
Modified version of the Hollander wound evaluation scale | 6 months follow up visit
  Includes several factors of cosmetic wound healing (skin puckering, patient satisfaction, etc.). Based on photographic and patient follow-up information
Modified version of the Hollander wound evaluation scale | 1 year follow up visit
  Includes several factors of cosmetic wound healing (skin puckering, patient satisfaction, etc.). Based on photographic and patient follow-up information

CONTACTS AND LOCATIONS:
Overall Officials: Chadi Tannoury, MD, Study Chair — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Denaro V, Di Martino A. Cervical spine surgery: an historical perspective. Clin Orthop Relat Res. 2011 Mar;469(3):639-48. doi: 10.1007/s11999-010-1752-3. PMID 21213087
- [Background] Fransen P. A simplified technique for anterior cervical discectomy and fusion using a screw-plate implanted over the Caspar distractor pins. Acta Orthop Belg. 2010 Aug;76(4):546-8. PMID 20973364
- [Background] Fehlings MG, Arvin B. Surgical management of cervical degenerative disease: the evidence related to indications, impact, and outcome. J Neurosurg Spine. 2009 Aug;11(2):97-100. doi: 10.3171/2009.5.SPINE09210. PMID 19769487